CLINICAL TRIAL: NCT07170956
Title: Variability in Tooth Root Number: A Cross-Sectional Study
Brief Title: Analysis of Tooth Root Number
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital of the Ministry of Interior, Kielce, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: CT/2025/1
Record Dates: First submitted 2025-09-04; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Tooth Abnormalities; Tooth Abnormality; Tooth Anatomy; Tooth Development Disorder; Tooth Disorder
Keywords: Tooth root; Tooth abnormalities; Tooth anatomy
MeSH Terms: conditions — Tooth Abnormalities; Tooth Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Females: Female patients
- Males: Male patients

SUMMARY:
The aim of this cross-sectional study is to assess the number of roots in permanent teeth. For this reason, researchers will conduct an analysis of CBCT scans. The collected data will be used for epidemiological analysis, including an examination of differences in outcomes between male and female patients.

DETAILED DESCRIPTION:
This study will involve analysis of anonymised CBCT images from Polish dental imaging facility. The analysis will include patients whose scans were obtained previously for diagnostic and therapeutic reasons and do not show significant artefacts. The primary outcome will be defined as the number of roots of each of the assessed teeth. Statistical analysis will be conducted in subgroups based on tooth type, patient gender, and patient age. This study has been approved by the bioethics committee.

ELIGIBILITY:
Inclusion Criteria:

* CBCT scans obtained following a written referral from a dentist,
* clear and complete visibility of the assessed structure,
* completed development of assessed roots.

Exclusion Criteria:

* incomplete root development in teeth other than third molars within the dentition,
* CBCT scans with significant artefacts.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General population of patients referred for CBCT for diagnostic or therapeutic reasons
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Tooth root number | The assessment is conducted once at the time of enrolment
  Number of separate roots of a single tooth, regardless of the level of division

SECONDARY OUTCOMES:
Male/female ratio | The assessment is conducted once at the time of data analysis
  Proportion of different numbers of roots in male and female
Age odds ratio | The assessment is conducted once at the time of analysis
  Odds ratio of different numbers of roots with a distinction based on age

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Maxillofacial Surgery, Hospital of the Ministry of Interior, Kielce, Poland

IPD SHARING:
Plan to Share IPD: Undecided